CLINICAL TRIAL: NCT06217302
Title: Effectiveness and Safety of Sotagliflozin in Slowing Kidney Function Decline in Persons With Type 1 Diabetes and Moderate to Severe Diabetic Kidney Disease
Brief Title: Sotagliflozin to Slow Kidney Function Decline in Persons With Type 1 Diabetes and Diabetic Kidney Disease
Acronym: SUGARNSALT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alessandro Doria (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); The Kidney Foundation of Canada (Other); The Cleveland Clinic (Other); University of Michigan (Other); University of Colorado, Denver (Other); Northwestern University (Other); Washington University School of Medicine (Other); State University of New York - Upstate Medical University (Other); Providence Medical Research Center (Other); Stanford University (Other); Montefiore Medical Center (Other); University of Toronto (Other); University Health Network, Toronto (Other); University of Calgary (Other); University of Alberta (Other); University of British Columbia (Other); Institut de Recherches Cliniques de Montreal (Other); LMC Diabetes & Endocrinology Ltd. (Other); Joslin Diabetes Center (Other); Lexicon Pharmaceuticals (Industry); DexCom, Inc. (Industry); University of Washington (Other); Breakthrough T1D (Other)
Responsible Party: Sponsor-Investigator, Alessandro Doria, Senior Investigator and Professor of Medicine, Joslin Diabetes Center
Organization: Joslin Diabetes Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STUDY00000249
Record Dates: First submitted 2024-01-09; First posted 2024-01-22 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Nephropathies; Kidney Failure, Chronic; Diabetes Mellitus Type 1; Heart Failure
Keywords: Diabetic Nephropathies; Kidney Failure, Chronic; Type 1 diabetes; Heart failure; Cardiovascular disease; Glomerular filtration rate; SGLT2 inhibitors; Diabetic kidney disease
MeSH Terms: conditions — Diabetic Nephropathies; Kidney Failure, Chronic; Diabetes Mellitus, Type 1; Heart Failure; Cardiovascular Diseases | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sotagliflozin (Active Comparator): Oral sotagliflozin at a dose of 200 mg (one tablet) per day for three years followed by a 2-month wash-out period.
  Interventions: Drug: Sotagliflozin
- Placebo (Placebo Comparator): Oral tablets similar to sotagliflozin tablets but containing no active drug (one tablet per day for three years followed by a 2-month wash-out period).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sotagliflozin — Oral sotagliflozin (200 mg per day)
  Other Names: INPEFA
  Arms: Sotagliflozin
Drug: Placebo — Inactive tablets identical to sotagliflozin tablets
  Arms: Placebo

SUMMARY:
Powerful new drugs that can prevent or delay end stage kidney disease (ESKD) - so called sodium-glucose cotransporter-2 inhibitors (SGLT2i) - are now available for patients with type 2 diabetes. Whether these drugs have similar effects in patients with type 1 diabetes (T1D) remains unknown because of the few studies in this population, due to concerns about the increase in risk of diabetic ketoacidosis (DKA, a serious, potentially fatal acute complication of diabetes due to the accumulation of substances called ketone bodies) observed with SGLT2i therapy in T1D. One of the few T1D studies conducted to date showed that implementing an enhanced DKA prevention plan can reduce the risk of DKA associated with the SGLT2i sotagliflozin (SOTA) to very low levels. In the present study, a similar DKA prevention program will be used to carry-out a 3-year trial to test the kidney benefit of SOTA in 150 persons with T1D and moderate to advanced DKD. After a 2-month period, during which diabetes care will be standardized and education on monitoring and minimizing DKA implemented, eligible study subjects will be randomly assigned (50/50) to take one tablet of SOTA (200 mg) or a similarly looking inactive tablet (placebo) every day for 3 years followed by 2-months without treatment. Neither the participants nor the study staff will know whether a person was assigned to taking SOTA or the inactive tablet. Kidney function at the end of the study will be compared between the two treatment groups to see whether SOTA prevented kidney function loss in those treated with this drug as compared to those who took the inactive tablet. The DKA prevention program will include participant education, close follow-up with study staff, continuous glucose monitoring, and systematic ketone body self-monitoring with a meter provided by the study. If successful, this study will provide efficacy and safety data that could be used to seek FDA approval of SOTA for the prevention of kidney function decline in patients with T1D and DKD.

DETAILED DESCRIPTION:
Despite improvements in glycemia management and the use of renin-angiotensin system blockade (RASB), the overall incidence of ESKD incidence in the US T1D population is not decreasing. For patients with type 2 diabetes (T2D), powerful new drugs that can prevent or delay ESKD, sodium-glucose cotransporter-2 inhibitors (SGLT2i), are now available. Whether similar results can be achieved in T1D remains unknown because of the paucity of studies in this population, due to concerns about the 2- to 3-fold increase in risk of diabetic ketoacidosis (DKA) associated with SGLT2i therapy in T1D. One of the few T1D studies conducted to date (inTandem, a sotagliflozin [SOTA] trial), showed that implementation of an enhanced DKA risk monitoring and mitigation strategy can reduce DKA incidence to <1%/year in subjects on 200 mg/day of this dual SGLT1 and SGLT2 inhibitor. The goals of the present study are to evaluate the renal effectiveness of SGLT2i in T1D and to better understand the benefit/risk ratio of SOTA in T1D persons with moderate to advanced diabetic kidney disease (DKD) - two goals that are warranted and critical given the high risk of death and ESKD in this population. The study, carried out by the Preventing Early Renal Loss (PERL) and the Canadian Institute of Health Research (CIHR)-funded SUGARNSALT (S&S) consortia, is a multi-center, double-blind, placebo-controlled, parallel-group randomized clinical trial in 150 patients with T1D and moderate to advanced diabetic kidney disease (estimated glomerular filtration rate [eGFR] 20-60 ml/min/1.73 m2 and ACR>200 mg/g). After a 2-month run-in period, during which diabetes care is standardized and education on monitoring and minimizing DKA implemented, eligible study subjects are randomized in a 1:1 ratio to receive placebo or once daily 200 mg SOTA for 3 years followed by a 2-month wash-out period. The eGFR at the end of the wash-out adjusted by its baseline value will be used as the primary outcome on which SOTA efficacy on DKD progression will be evaluated. An intensive DKA risk mitigation plan will be implemented based on the inTandem enhanced protocol as well as on the STICH (Stop SGLT2i, Insulin administration, Carbohydrate intake, Hydration) and STOP-DKA protocols. Cornerstones of this plan will be enhanced participant education, close follow-up with study staff, continuous glucose monitoring, and systematic ketone body (beta-hydroxybutyrate [BHB]) self-monitoring. If successful, the present study will provide efficacy and safety data that could be used to seek FDA and Health Canada approval of SOTA for a T1D DKD indication. Based on the available data in T1D, it can be conservatively postulated that SOTA may reduce eGFR loss by 2 ml/min/1.73 m2 per year. Depending on the baseline eGFR, this would translate to a 5-10 year delay of ESKD. The reduction in morbidity and mortality resulting from the prevention or delay of ESKD due to the use of SOTA would have a major impact on the lives of T1D patients with significant DKD as well as on society at large, substantially reducing the human and financial costs associated with this condition.

ELIGIBILITY:
Inclusion Criteria:

* Type1 diabetes (T1D) continuously treated with insulin within one year from diagnosis.
* Duration of T1D ≥ 8 years;
* eGFR based on serum creatinine and cystatin c (2021 serum creatinine-cystatin C CKD-EPI equation) between 20 and 60 ml/min/1.73 m2 at screening (with the option of a second eGFR measurement within 4 weeks from the first one if the eGFR was in the range of >60 to ≤65 or ≥16 to <20 ml/min/1.73 m2);
* a. First morning void urinary albumin creatinine ratio (UACR) ≥200 mg/g at Screening or on repeat measurement within 4 weeks from the first one, or b. First morning void urinary UACR ≥100 mg/g at Screening or on repeat measurement within 4 weeks and at least one uACR >=30 in the previous 2 years while treated with RASB at a stable dose;
* HbA1c at screening <10% (with the option of a second HbA1c measurement within 4 weeks from the first one if the HbA1c was ≤10.2%);
* Receiving standard of care, including renin angiotensin system blockers (RASB) at a clinically appropriate dose, unless contraindicated or not tolerated.
* Willing and able to comply with schedule of events and protocol requirements, including written informed consent, and willing to wear a continuous glucose monitoring (CGM) device for the entire duration of the study.
* a. Blood pressure ≤155/95 mmHg at screening, or b. BP ≤155/95 mmHg at the end of the run-in period, or c. consistent BP ≤155/95 mmHg on home monitoring during the run-in period, as determined by study site investigator, despite BP values >155/95 mmHg in clinic.

Exclusion Criteria:

* Type 2 diabetes or monogenic forms of diabetes or diabetes secondary to pancreatic disease;
* Use of automated insulin delivery devices that are not approved by health regulatory agencies, or used in ways that do not align with manufacturer recommendations;
* Use of any SGLT inhibitor in the previous 2 months;
* Use of dual medication RASB therapy (spironolactone, eplerenone, finerenone are allowed in combination with RASB therapy);
* Use of GLP-1 receptor agonists and other non-insulin glucose-lowering agents if not on stable dose for > 2 months at screening (patients can be rescreened after being on stable dose for > 2 months);
* Use of anti tumor necrosis factor (TNF) alpha biologic medications at screening;
* Known allergies, hypersensitivity, or intolerance to SOTA;
* History of ≥3 severe hypoglycemic events (requiring third-party assistance for correction) within 3 months of screening;
* History of diabetic ketoacidosis (DKA) or non-ketotic hyperosmolar state within 3 months of screening OR >1 episode of DKA or non-ketotic hyperosmolar state within 12 months of screening;
* Blood beta-hydroxybutyrate (BHB) >0.6 mmol/L for >2 hours on >2 occasions during the Run-in period;
* Inadequate beta hydroxybutyrate (BHB) testing (<50% of the prescribed measurements) during Run-in;
* History of primary renal glycosuria;
* History of biopsy-proven non-diabetic chronic kidney disease (CKD);
* History of kidney transplant or currently on chronic dialysis;
* Current or past history of decompensated cirrhosis (defined as variceal bleeding, ascites or hepatic encephalopathy), and/or known diagnosis of cirrhosis based on liver biopsy, imaging, or elastography, and/or aspartate aminotransferase (AST) or alanine transaminase (ALT) at screening >2 times upper limit of normal, and/or total bilirubin at screening >1.3 times upper limit of normal).
* History of severe acquired immune deficiency syndrome or human immunodeficiency virus (HIV) infection or severely immunocompromised status;
* Cancer treatment (excluding non-melanoma skin cancer treated by excision, carcinoma in situ of the cervix or uterus, ductal breast cancer in situ, resected non-metastatic breast or prostate cancer) within one year of screening.
* Illicit drug abuse within 6 months of screening;
* Heavy alcohol use (for men, 5 drinks or more on any day or 15 drinks or more per week; for women, 4 drinks or more on any day or 8 drinks or more per week);
* Participation in another interventional clinical research study within 30 days of screening;
* Breastfeeding, pregnancy, or unwillingness to be on contraception during the trial;
* Presence of a clinically significant medical history, physical examination, or laboratory finding that may interfere with any aspect of study conduct or interpretation of results;
* Any condition that may render the patient unable to comply with study requirements and/or complete the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
eGFR at the end of the wash-out period following the treatment period | End of the 2-month wash-out period following the 3-year treatment period (weeks 162 and 164)
  eGFR at the end of the 8-week drug washout period following the 3-year treatment period, estimated from Central Lab serum creatinine and cystatin C using the 2021 Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation and adjusted by its baseline value. Baseline and end-of-washout eGFRs will be considered as the average of two eGFR values taken on two separate days before randomization (V2 and V4) and after the washout (V18 and V19), respectively.

SECONDARY OUTCOMES:
Time to ≥40% eGFR decline from baseline, kidney failure , or death from renal causes | Up to the end of the 2-month wash-out period following the 3-year treatment period (week 0 to 164)
  Time from randomization to 1. sustained ≥40% eGFR decline (based on eGFR estimated from serum creatinine and cystatin C using the 2021 CKD-EPI equation) confirmed after 30 days; 2. kidney failure, defined by eGFR ≤10ml/min/ 1.73m2 confirmed after 30 days or occurring within 30 days prior to death, or initiation of maintenance kidney replacement therapy; or 3. death from kidney-related causes. If an eGFR value meeting the above criteria is observed at the last study visit or immediately before a participant is lost to follow-up or withdraws from the study, no confirmation of this value will be necessary.

OTHER OUTCOMES:
eGFR at the end of the 3-yr treatment period | End of the 3-year treatment period (week 156)
  eGFR at the end of the 3-yr treatment period (before the washout period) adjusted for the baseline value
Time to fatal or non-fatal cardiovascular disease (CVD) events | Up to the end of the 2-month wash-out period following the 3-year treatment period (week 0 to 164)
  Time to fatal or non-fatal CVD events (CV death, non-fatal myocardial infarction, non-fatal stroke, or coronary, carotid, or peripheral revascularization procedures)
Time to hospitalization or urgent visit for heart failure or CV death | Up to the end of the 2-month wash-out period following the 3-year treatment period (week 0 to 164)
  Time to hospitalization or urgent visit for heart failure or death for cardiovascular causes
Time to hospitalization for heart failure | Up to the end of the 2-month wash-out period following the 3-year treatment period (week 0 to 164)
  Time to hospitalization for heart failure
B-type natriuretic peptide (NTproBNP) serum levels at the end of the drug washout | End of the 2-month wash-out period following the 3-year treatment period (week 164)
  Serum levels of NTproBNP at the end of the 8-week drug washout, adjusted for its baseline value
High-sensitivity cardiac troponin (hs-cTnT) serum levels at the end of the drug washout | End of the 2-month wash-out period following the 3-year treatment period (week 164)
  Serum levels of hs-cTnT at the end of the 8-week drug washout, adjusted for its baseline value
NTproBNP serum levels at the end of the treatment period | End of the 3-year treatment period (week 156)
  Serum levels of B-type natriuretic peptide (NTproBNP) at the end of the 3-year treatment period, adjusted for its baseline value
hs-cTnT serum levels at the end of the treatment period | End of the 3-year treatment period (week 156)
  Serum levels of high-sensitivity cardiac troponin (hs-cTnT ) at the end of the 3-year treatment period, adjusted for its baseline value
Mean blood HbA1c levels during the treatment period | Weeks 0, 2, 8, 16, 28, 44, 60, 76, 92, 108, 124, 140 156 (from baseline to the end of the treatment period)
  Mean HbA1c during the 3-year treatment period
Mean blood glucose levels during the treatment period | Weeks 2, 8, 16, 28, 44, 60, 76, 92, 108, 124, 140 156 (from baseline to the end of the treatment period)
  Mean blood glucose from continuous glucose monitoring during the 3-year treatment period
Mean GMI during the treatment period | Weeks 2, 8, 16, 28, 44, 60, 76, 92, 108, 124, 140 156 (from baseline to the end of the treatment period)
  Mean glucose management indicator (GMI) from continuous glucose monitoring during the 3-year treatment period
Mean time in range (TIR) during the treatment period | Weeks 2, 8, 16, 28, 44, 60, 76, 92, 108, 124, 140 156 (from baseline to the end of the treatment period)
  Mean time with blood glucose in the 70 to 180 mg /dl range from continuous glucose monitoring during the 3-year treatment period
Mean time below range 70 (TBR70) during the treatment period | Weeks 2, 8, 16, 28, 44, 60, 76, 92, 108, 124, 140 156 (from baseline to the end of the treatment period)
  Mean time with blood glucose below 70 mg/dl from continuous glucose monitoring during the 3-year treatment period
Mean time below range 54 (TBR54) during the treatment period | Weeks 2, 8, 16, 28, 44, 60, 76, 92, 108, 124, 140 156 (from baseline to the end of the treatment period)
  Mean time with blood glucose below 54 mg/dl from continuous glucose monitoring during the 3-year treatment period
Mean time above range 180 (TAR180) during the treatment period | Weeks 2, 8, 16, 28, 44, 60, 76, 92, 108, 124, 140 156 (from baseline to the end of the treatment period)
  Mean time with blood glucose above 180 mg/dl from continuous glucose monitoring during the 3-year treatment period
Mean time above range 250 (TAR250) during the treatment period | Weeks 2, 8, 16, 28, 44, 60, 76, 92, 108, 124, 140 156 (from baseline to the end of the treatment period)
  Mean time with blood glucose above 250 mg/dl from continuous glucose monitoring during the 3-year treatment period
Mean Glucose CV during the treatment period | Weeks 2, 8, 16, 28, 44, 60, 76, 92, 108, 124, 140 156 (from baseline to the end of the treatment period)
  Mean blood glucose coefficient of variation (CV) from continuous glucose monitoring during the 3-year treatment period
Mean MAGE during the treatment period | Weeks 2, 8, 16, 28, 44, 60, 76, 92, 108, 124, 140 156 (from baseline to the end of the treatment period)
  Mean amplitude of glycemic excursions (MAGE) from continuous glucose monitoring during the 3-year treatment period
Mean GRI during the treatment period | Weeks 2, 8, 16, 28, 44, 60, 76, 92, 108, 124, 140 156 (from baseline to the end of the treatment period)
  Mean glycemic risk index (GRI) from continuous glucose monitoring during the 3-year treatment period
Mean total daily insulin dose during the treatment period | Weeks 2, 8, 16, 28, 44, 60, 76, 92, 108, 124, 140 156 (from baseline to the end of the treatment period)
  Mean total daily insulin dose (TDD, units/kg) during the 3-year treatment period
Urinary albumin excretion rate change from baseline equal to or more negative than -30% at the end of treatment | End of treatment period (Week 156).
  Urinary albumin excretion rate (UAER, timed overnight collection) reduction from baseline ≥30% at the end of treatment;
Urinary albumin excretion rate change from baseline equal to or more negative than -30% at the end of the washout period | End of the 2-month wash-out period following the 3-year treatment period (week 164)
  Urinary albumin excretion rate (UAER) reduction from baseline ≥30% at the end of the 8-week washout period following the 3-year treatment period;
eGFR slope during the treatment period | Weeks 0, 2, 8, 16, 28, 44, 60, 76, 92, 108, 124, 140 156 (from baseline to the end of the treatment period)
  eGFR slope from baseline to the end of the 3-yr treatment period (before the washout period), kidney failure, death, or study discontinuation, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Doria, MD PhD MPH, Principal Investigator — Joslin Diabetes Center; Michael Mauer, MD, Principal Investigator — University of Minnesota; David Cherney, MD PhD, Principal Investigator — University of Toronto
Locations (18):
- United States (12):
  - Stanford University Medical Center, Stanford, California
  - Barbara Davis Center / University of Colorado Denver, Aurora, Colorado
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Joslin Diabetes Center, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - SUNY Upstate Medical University, Syracuse, New York
  - Albert Einstein College of Medicine / Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Texas Southwestern, Dallas, Texas
  - University of Washington, Seattle, Washington
  - Providence Sacred Heart Medical Center, Spokane, Washington
- Canada (6):
  - Unversity of Calgary, Calgary, Alberta
  - Alberta Diabetes Institute, Edmonton, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - LMC Diabetes and Endocrinology, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Institut de Recherches Cliniques de Montréal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Raalte DH, Bjornstad P, Persson F, Powell DR, de Cassia Castro R, Wang PS, Liu M, Heerspink HJL, Cherney D. The Impact of Sotagliflozin on Renal Function, Albuminuria, Blood Pressure, and Hematocrit in Adults With Type 1 Diabetes. Diabetes Care. 2019 Oct;42(10):1921-1929. doi: 10.2337/dc19-0937. Epub 2019 Aug 1. PMID 31371432
- [Background] Bhatt DL, Szarek M, Pitt B, Cannon CP, Leiter LA, McGuire DK, Lewis JB, Riddle MC, Inzucchi SE, Kosiborod MN, Cherney DZI, Dwyer JP, Scirica BM, Bailey CJ, Diaz R, Ray KK, Udell JA, Lopes RD, Lapuerta P, Steg PG; SCORED Investigators. Sotagliflozin in Patients with Diabetes and Chronic Kidney Disease. N Engl J Med. 2021 Jan 14;384(2):129-139. doi: 10.1056/NEJMoa2030186. Epub 2020 Nov 16. PMID 33200891
- [Background] Bhatt DL, Szarek M, Steg PG, Cannon CP, Leiter LA, McGuire DK, Lewis JB, Riddle MC, Voors AA, Metra M, Lund LH, Komajda M, Testani JM, Wilcox CS, Ponikowski P, Lopes RD, Verma S, Lapuerta P, Pitt B; SOLOIST-WHF Trial Investigators. Sotagliflozin in Patients with Diabetes and Recent Worsening Heart Failure. N Engl J Med. 2021 Jan 14;384(2):117-128. doi: 10.1056/NEJMoa2030183. Epub 2020 Nov 16. PMID 33200892
- [Background] Markham A, Keam SJ. Sotagliflozin: First Global Approval. Drugs. 2019 Jun;79(9):1023-1029. doi: 10.1007/s40265-019-01146-5. PMID 31172412
- [Derived] Nardone M, Kugathasan L, Sridhar VS, Dutta P, Campbell DJT, Layton AT, Perkins BA, Barbour S, Lam TKT, Levin A, Lovblom LE, Mucsi I, Rabasa-Lhoret R, Rac VE, Senior P, Sigal RJ, Stanimirovic A, Persson F, Stougaard EB, Doria A, Cherney DZI. Modeling Cardiorenal Protection with Sodium-Glucose Cotransporter 2 Inhibition in Type 1 Diabetes: An Analysis of DEPICT-1 and DEPICT-2. Clin J Am Soc Nephrol. 2025 Apr 1;20(4):529-538. doi: 10.2215/CJN.0000000641. Epub 2025 Feb 7. PMID 39918875